

# AI 辅助胃镜下静脉曲张诊断的前瞻性多中 心研究

## 研究方案

**项目负责人:** 陈明锴 消化内科 13720330580

**项目联系人:** 肖勇 消化内科 13886150643

柯舸 消化内科 18296376562

版本号: V 4.0 , 版本日期: 2021-11-08





## AI 辅助胃镜下静脉曲张诊断的前瞻性多中心研究

简称: AI-assisted diagnosis research

| 方案版本 | 4.0 |
|-------|--------------------------------|
| 版本日期 | November 08,2021 |
| 国家 | ■ 中国 |
| 研究产品 | Artificial Intelligence |
| 主要研究者 | 陈明锴 教授 |
| 地址 | 湖北武汉武昌区张之洞路(原紫阳路)99 号解放路 238 号 |

本方案属于武汉大学人民医院,本方案中包含的信息是保密的,仅供参与临床试验的相 关方使用,未经允许不得对外披露。



## 目录

| 1. | 概要 | | | 4 |
|----|-------|-------------|-----------|-----|
| | 1.1. | 时间和 | 1事件表 | 6 |
| | 1.2. | 研究流 | [程图 | 7 |
| 2. | 介绍 | | | 8 |
| 3. | 受试者 | 皆的定义 | <u></u> | 8 |
| | 3. 1. | 入选标 | ·准 | 8 |
| | 3. 2. | 排除标 | 术 | 9 |
| | 3. 3. | 受试者 | 行入组的定义 | 9 |
| 4. | 终点占 | ラ假设 | | 9 |
| | 4.1. | 主要终 | 3点 | 9 |
| | 4.2. | 次要终 | 3点 | 9 |
| 5. | 研究目 | 目的与总 | .体设计 | 10 |
| | 5. 1. | 研究目 | 的 | 10 |
| | 5. 2. | 总体设 | <u></u> ት | 10 |
| 6. | 研究》 | <b>沧程</b> | | 10 |
| | 6.1. | 研究流 | 冠程总体概述 | 10 |
| | 6.2. | 受试者 | 行入组 | 10 |
| | 6 | . 2. 1. | 受试者知情同意书 | 10 |
| | 6 | . 2. 2. | 受试者筛选 | 11 |
| | 6 | . 2. 3. | 受试者识别编号 | 11 |
| | 6.3. | 试验干 | -预流程 | 11 |
| | 6.4. | 中止与 | 5退出 | 11 |
| 7. | 方案制 | 削定依据 | 号与风险/获益分析 | 12 |
| | 7. 1. | 研究总 | .体设计方法 | 12 |
| | 7. 2. | 评价终 | · 点选择 | 12 |
| | 7. 3. | 研究人 | 、群的界定 | 12 |
| | 7.4. | 相关受 | · 益 | 12 |
| | 7. 5. | 整体可 | 「行性分析 | 12 |
| 8. | 数据管 | <b>曾理与统</b> | 计分析 | 13 |
| | 8.1. | 数据管 | 7理与统计分析计划 | 13 |
| | 8.2. | 统计方 | ī法 | 13 |
| | 8.3. | 假设检 | 39金 | 13 |
| | 8.4. | 样本量 | 也的计算 | 13 |
| 9. | 关于和 | 斗研门诊 | 意见的回答 | 14 |
| 10 | 会老で | ナ武 | | 1.4 |



## 1. 概要

| 标题: | AI 辅助胃镜下静脉曲张诊断的前瞻性多 |
|-------|-----------------------------------------|
| | 中心研究 |
| 简称: | AI improving diagnostic research |
| 研究产品: | Artificial intelligence |
| 主要终点: | AI 对食管胃静脉曲张诊断及内镜下表现 |
| | (形式、颜色、红色征、出血征和黏膜表 |
| | 现)描述和治疗建议的准确度 |
| 次要终点 | (1) 与参考标准相比, AI 和第三方医生给 |
| | 出诊断的准确度、特异度、灵敏度 |
| | (2) 与参考标准相比, AI 和第三方医生对 |
| | 患者危险度的判断准确度(根据专家 |
| | 意见将患者分为高危、低危患者,分 |
| | 别统计准确度) |
| | (3) 与参考标准相比 AI 和第三方医生提 |
| | 出治疗建议的准确度 |
| | (4) 回归分析各项诊断指标对食管胃静 |
| | 脉曲张的危险影响程度,并评估 AI |
| | 在重要诊断指标上的准确度 |
| | (5) 第三方医师在 AI 辅助下,对之前诊 |
| | 断有差异的视频的纠错率 |
| 研究设计: | <b>党设计:</b> 多中心、对照 |
| | 01 尹河十兴 星医院 09 复日十兴中山医院 02 米江十兴医兴院附居签 |
| 研究中心 | 01 武汉大学人民医院、02 复旦大学中山医院、03 浙江大学医学院附属第 |
| ካሊተኄ | 一医院、04 山西煤炭总医院、05 新疆医科大学附属第一医院、06 西南医 |
| | 院、07 宜昌市中心医院、08 恩施州中心医院、09 孝感第一医院、10 普仁 |
| | 医院、11 阜阳市第二医院 |
| 受试人群: | 2022年1月至2022年12月于本研究各中心就诊的肝硬化患者及第三方 |
| | 医师 |
| 样本量: | 预计纳入肝硬化患者 793 例, 医师数量 23 位 |
| 研究流程: | 本研究为多中心前瞻性研究,符合研究纳入排除标准的患者,于门诊及住 |
| | 院期间收集其基本信息,由指定医生向患者介绍此次研究的意义并签署知 |
| | 情同意书。在患者内镜检查结束后,收集保存内镜下操作视频,导入AI |



得到其对上述特征的结论以及分层和治疗建议。后续要求符合纳入标准的第三方医师,记录其观看视频后得出的各项诊疗建议(主要以选择问卷形式,避免主观上的偏差),问卷内容包括其在内镜操作视频中观察到的静脉曲张相关特征(有无红色征、出血征,曲张静脉的形态、直径、颜色、黏膜征),同时要求给出相应危险分层及治疗建议。对 AI 与医师得出不一致结论的视频,将让医师再次观看带有 AI 提示的这些视频给出意见,首次与再次观看之间将会有两周的缓冲期。诊断的参考标准将会由三名内镜专家各自观看不带 AI 提示的视频得出,以三名专家得出的结论为参考标准,当三名专家具有不一致的结论时,以三者讨论得出一致意见为准,若最终无法达成一致,弃用该视频。

通过对医师以及 AI 给出诊断的准确度对比来获得主要及次要终点。所有数据采用 SPSS 统计软件完成统计分析。

安全性:

本试验仅涉及与诊断相关的研究, 可以保证安全性



## 1.1. 时间和事件表

| 内镜医师 | 内镜前 | 内镜后 |
|----------|-----|-----|
| 知情同意 | X | |
| 年龄 | X | |
| 性别 | X | |
| 学历 | X | |
| 执业年数 | X | |
| 内镜操作年数 | X | |
| 操作胃镜数量 | X | |
| 接触静脉曲张年数 | X | |
| 纠错率 | | X |
| 诊断表 | | X |

| 患者 | 内镜前 | 内镜后 |
|------|-----|-----|
| 知情同意 | X | |
| 年龄 | X | |
| 性别 | X | |
| 身份信息 | X | |
| 联系方式 | X | |



## 1.2. 研究流程图





## 2. 介绍

食管胃静脉曲张破裂出血(esophagogastric variceal bleeding, EGVB)是肝硬化失代偿期门静脉高压最常见的并发症之一,大约 50%的肝硬化患者存在食管胃静脉曲张,一旦发展为静脉曲张破裂出血,六周死亡率达 25%【1-4】,因此高出血风险的肝硬化患者的一级预防尤为重要。

虽然门脉高压是导致食管胃底静脉曲张的直接原因,但诊断以肝静脉压力梯度测定为标准,该操作受限于设备以及较高的费用,不适于广泛应用。各类肝硬化指南也指出定期的内镜检查有助于肝硬化患者出血事件的预防与控制,但内镜检查的结论准确度依赖临床医师的经验,主观占比较大,为提高内镜医师对食管胃静脉曲张筛查的工作效率和诊断准确率,我们亟需一款能提供实时、高效、客观诊断建议的智能系统。

多项研究已对食管胃静脉曲张的内镜下表现进行了危险分成,主要包括有无红色征、出血征,曲张静脉的形态、直径、颜色、黏膜征。AI基于上述危险因素,采用深度卷积神经网络(DNCC)对获得的肝硬化患者食管胃静脉曲张视频及图像自动分层学习,已初步构建完成相关预测模型,并以人机大赛方式检测其准确性,结果证明 AI 确实能提高实时过程中预测食管胃静脉曲张的风险因素的效率和准确性【5】。

## 3. 受试者的定义

患者: 2022年1月至2022年12月于本研究各中心就诊的肝硬化患者。

内镜医师:符合内镜医师纳入标准的第三方内镜医师。

#### 3.1. 入选标准

#### 符合以下具体标准的患者将被考虑纳入本研究:

- 1) 年龄在18岁(含)以上的男性或女性;
- 2) 需要进行胃镜及其相关检查进一步明确消化道疾病特征;
- 3) 肝硬化患者,有门静脉高压的体征或症状,有进行内镜检查筛查静脉曲张的临床指征。
- 4) 能够阅读、理解并签署知情同意书;
- 5) 研究者认为受试者能够理解该临床研究的流程,愿意并能够完成所有的研究程序和 随访访视,配合研究程序;

#### 符合以下具体标准的内镜医师将被考虑纳入本研究:

- 1) 从事内镜相关工作的医师
- 2) 具备良好的研究态度,充分理解病例报告表中各项指标的含义
- 3) 能够阅读、理解并签署知情同意书



### 3.2. 排除标准

#### 符合以下任一具体标准的患者将被拒绝参与本研究:

- 1) 孕期或哺乳期妇女;
- 2) 既往食管胃外科手术史的患者;
- 3) 既往接受过介入或内镜下处理的患者:
- 4) 患者存在不适宜参加临床试验的高危疾病或其它特殊情况;
- 5) 患者明确诊断有食管或胃部憩室、息肉、癌等可能影响静脉曲张观察的疾病;
- 6) 患者内镜视频经三位专家观看后无法达成一致诊疗意见。

#### 符合以下任一具体标准的医师将被拒绝参与本研究:

- 1) 未接触或极少接触肝硬化病人检查的内镜医师
- 2) 不宜参加研究的其他情况

## 3.3. 受试者入组的定义

患者受试者在经研究者评估后确认符合纳排标准并签署知情同意书后且即入组, 医师受试者符合纳排标准并签署知情同意书即入组。

## 4. 终点与假设

## 4.1. 主要终点

AI 对食管胃静脉曲张诊断及内镜下表现(形式、颜色、红色征、出血征和黏膜表现)描述和治疗建议的准确度。

#### 4.2. 次要终点

- (1) 与参考标准相比, AI 和第三方医师给出诊断的准确度、特异度、灵敏度
- (2) 与参考标准相比,AI 和第三方医师对患者危险度的判断准确度(根据专家意见将患者分为高危、低危患者,分别统计准确度)
- (3) 与参考标准相比 AI 和第三方医师提出治疗建议的准确度
- (4) 回归分析各项诊断指标对食管胃静脉曲张的危险影响程度,并评估 AI 在重要诊断指标上的准确度
- (5) 第三方医师在 AI 辅助下,对之前诊断有差异的视频的纠错率



## 5. 研究目的与总体设计

#### 5.1. 研究目的

通本研究主要是验证 AI 建立的食管胃静脉曲张诊断模型的临床准确性

### 5.2. 总体设计

本研究为一项前瞻性、多中心、开放性的临床研究。该研究共在 11 个中心进行,预计入组793例患者,23 位内镜医师

#### 6. 研究流程

## 6.1. 研究流程总体概述

- 签署知情同意书
- 受试者基础资料的收集
- 获取内镜操作视频
- 各中心严格按纳排标准入组医师及患者
- 按主要及次要终点分别获取专家、医师、AI 的诊断意见
- 计算获得主要及次要终点

#### 6.2. 受试者入组

受试者签署知情同意书后,方可完成研究相关资料收集及与本研究相关的测试。

### 6.2.1. 受试者知情同意书

根据赫尔辛基宣言,在未提供充分的知情同意情况下不允许受试者参加研究。主要研究 者负责确保在没有提供充分的知情同意情况下,没有受试者入选研究。未能获得知情同 意且未正确记录此流程视为违反了赫尔辛基宣言和本研究方案。

所有知情同意文件(ICD)必须获得伦理的支持。受试者的知情同意需要受试者本人并以受试者的主要语言在知情同意文件上记录。

受试者需进行初步筛选,以确定其是否大体符合研究的资格标准。如果满足,签署知情同意书后则认为其以被纳入研究。在签署知情同意书之前,研究者或经过适当培训的指



定人员应确认受试者理解研究中的以下各点:

- 研究的目的,
- 带来的潜在风险或不良事件,
- 与参与研究直接相关的潜在风险或不良事件,
- 研究的要求包括随访访视,
- 受试者作为临床研究参与者的所有权利。

在对研究目的进行解释之后,研究者或经过培训的指定人员应回答受试者的任何问题。如果受试者同意参与,他或她的意愿必须通过在 EC 批准的 ICF 上签名和注明日期进行记录,并且该文件由获得知情同意的人签署并注明日期。

成功完成知情同意过程后, 研究者或经培训的指定人员将根据研究需要对受试者进行随机分组。

## 6.2.2. 受试者筛选

对在各中心接诊的肝硬化患者及从事内镜工作的医师根据入排标准进行筛选,满足筛选标准的患者及医师受试者入组。为证实受试者的选择不存在偏移,筛选的日期、结果(是否入组)和受试者未入选的主要原因(例如,不符合入排标准、没有兴趣参加研究)将存在该记录中。患者的入组将在各中心采用竞争入组的方式,达到预期数量后研究结束,患者入组后,研究中心将要完成研究数据收集。

#### 6.2.3. 受试者识别编号

在获得知情同意后对受试者进行编号。

患者受试者编号以 PS 作为固定开头,以研究中心编号作为首位数字,如武汉大学人民 医院为 01,依获得知情同意书的时间从 001 开始编号。例如武汉大学人民医院的第 1 位签署知情同意书的受试者编号为 PS01001,其后第 2 位 PS01002。研究中心编号见研 究中心列表。医师受试者编号以 DS 作为固定开头,依获得知情同意书的时间从 001 开始编号。一旦分配受试者标识号后,该号便不可重复使用。

#### 6.3. 试验干预流程

本研究在受试者签署知情同意书后未进行任何干预措施。

#### 6.4. 中止与退出

受试者经筛选后确认符合参加该研究的资格、签署知情同意书并完成随机后则视为入组。若研究过程中受试者因主观或客观因素无法继续进行该项研究,退出研究的原因将被记录,退出受试者的编号将被保留,不会被替代,退出前的研究数据仍被纳入研究相关分析中。



## 7. 方案制定依据与风险/获益分析

使用 AI 对内镜检查提供辅助诊疗信息,该信息不会作为最终的诊断,患者所获得的诊疗仍是来自操作医师及临床医师,医师受试者在 AI 提供静脉曲张各个指标和总体风险评估等方面提示的基础上,自主作出应有的诊断。整个研究流程并不会影响到患者院内的诊疗,对受试者产生风险。

#### 7.1. 研究总体设计方法

<u>对照</u>: AI 和参考标准对同一份内镜视频材料的诊疗意见,参考标准为对照组; AI 和第三方医师对同一份内镜视频材料给出的诊疗意见,两者互为对照; 内镜医师在有无 AI 提示下对同一份视频材料给出的诊疗意见,为自身对照。

## 7.2. 评价终点选择

主要终点为 AI 对食管胃静脉曲张诊断及内镜下表现(形式、颜色、红色征、出血征和黏膜表现)描述和治疗建议的准确度:在参考标准下,以 AI 给出的正确的诊断与描述和治疗建议数目为分子,除以所有患者的数目。

参考标准:三名内镜方面的专家得出的一致诊断结论,若有一名专家诊断意见出现差异,则弃用该视频。

### 7.3. 研究人群的界定

患者受试者的纳入主要来自各中心就诊的肝硬化患者,在最低纳入数量的基础上,为了 尽量证实 AI 的准确度,尽可能多的纳入患者,但仍严格按纳排标准。

医师受试者的纳入主要来自已从业的内镜医师,为保证医师能较好的完成病例报告表的填写,研究过程中将为参与医师充分介绍研究的流程及注意事项,同时监督医师的完成进度及病例报告表完成度。

#### 7.4. 相关受益

患者受试者的内镜表现将由专家、AI、第三方医师共同进行诊断,一部分内镜表现复杂的患者将从中获益。医师受试者可在该研究过程中提高自身的内镜诊疗水平。

#### 7.5. 整体可行性分析

前期在武汉大学人民医院的其他试验中已经使用了 AI 相关数据集,整体可操作性较强。 同时 AI 诊断食管胃底静脉曲张的大样本回顾性研究已经完成。



## 8. 数据管理与统计分析

## 8.1. 数据管理与统计分析计划

数据管理与统计分析由武汉大学人民医院负责实施。

#### 8.2. 统计方法

本研究主要验证 AI 的准确率,以及 AI 与医师之间的差异性,大部分为计数资料,主要以频数(百分比)形式表示,组间比较采用卡方检验,必要时采用 Fisher 检验,所有分析均在预期 5%的双侧显著性上进行评估。

#### 8.3. 假设检验

主要有效性终点是 AI 对静脉曲张的诊断准确度与现在临床医生的平均诊断准确度相比 具有更优性或非劣效性。

主要终点的统计假设如下:

HO:PA-PB<0

H1:PA-PB≥0

PA, PB 分别为 AI 与医师受试者的诊断准确度。

当 PA 与 PB 均超过有效性介值且 PA≥PB, 拒绝 HO, 接受 H1。

#### 8.4. 样本量的计算

根据主要终点指标食管静脉曲张及其内镜下表现的总精度进行样本量预估,为单组临床试验,对于样本量测定,预期双侧显著性水平 5% ( $\alpha=5\%$ ),检验效能 power=80% ( $\beta=0.2$ ),脱落率 10%。以前期研究内镜下评估的精度进行样本量估算,估计 AI 的准确度 P=97%,医师准确率 93.94%,计算得到需要纳入肝硬化患者 793 人。

医师受试者的数量由于现在尚缺乏大量相关文献的报道,因此根据前期回顾性研究,医生的准确率 93.94%,采用抽样模拟,允许误差 10%,预期双侧显著性水平 5%,预计纳入 23 名医师。



## 9. 关于科研门诊意见的回答

- 1) 对于 AI 的准确性的判定:每份内镜视频,均会由三位专家观看后得到一致结论, 结论以递交的病例报告表形式呈现,每个观察指标均有明确的参考标准,而本研究 认定 AI 诊断正确的标准即是对表中的每一项指标,AI 给出的结论与专家的参考标 准都一致,若有一项于专家意见不同,即判定 AI 诊断错误。
- 2) 对于 AI 于第三方医师, 医师在有无 AI 辅助下的诊断意见的比较, 从研究目的出发, 对于 AI 于第三方医师的比较, 首要是比较两者诊断静脉曲张的准确度, 来说明 AI 在诊断方面是否优于内镜医师, 同时也会比较 AI 和第三方医师在每个指标上的准确度差异, 为进一步优化 AI 的诊断水平提供建议; 对于医师在有无 AI 提示下的诊断意见的比较, 从研究目的出发, 更多的是为了获得医生前后两次观看后是否能在 AI 的提示下对之前诊断有误的内镜视频达到纠正的效果, 在本研究中, 医生达到纠错的准则为只要对某一指标达到纠错的效果, 即认为 AI 对医师有所帮助, 因此在统计纠错率上主要会以单个指标的纠错率来进行统计, 同时兼顾总体静脉曲张的诊断纠错率。
- 3) 对于医师数量的计算,感谢科研门诊专家的指导,已按要求进行统计学修改。

## 10. 参考文献

- [1] EASL Clinical Practice Guidelines for the management of patients with decompensated cirrhosis. Journal of hepatology 69, 406-460 (2018).
- 【2】中华医学会肝病学分会,中华医学会消化病学分会,中华医学会内镜学分会,肝硬化门静脉高压食管胃静脉曲张出血的防治指南 Journal of Clinical Hepatology. 32, 203-219 (2016).
- [3] R. de Franchis, Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. Journal of hepatology 63, 743-752 (2015).
- [4] J. G. Karstensen et al., Endoscopic treatment of variceal upper gastrointestinal bleeding: European Society of Gastrointestinal Endoscopy (ESGE) Cascade Guideline. Endoscopy international open 8, E990-E997 (2020).
- [5] Mingkai Chen et al. Automated and real-time validation of gastroesophageal varices under esophagogastroduodenoscopy using deep convolutional neural network: a multicenter retrospective study (with video)[J]. Gastrointestinal Endoscopy, 2020.



| 姓名 | 职称 | 科室 | 项目分工 | 签名 |
|-----|----------|------|------------|----|
| 陈明锴 | 主任医师, 教授 | 消化内科 | 项目负责人 | |
| 肖勇 | 副主任医师 | 消化内科 | 项目联系人,质量控制 | |
| 柯舸 | 硕士研究生 | 消化内科 | 项目联系人,论文撰写 | |
| 曹卓 | 主治医师 | 消化内科 | 数据管理 | |
| 黄子殷 | 硕士研究生 | 消化内科 | 资料收集 | |
| 何安玲 | 硕士研究生 | 消化内科 | 资料收集 | |
| 刘小娇 | 硕士研究生 | 消化内科 | 资料收集 | |
| 邬海燕 | 硕士研究生 | 消化内科 | 资料收集 | |

签名:

日期: 年 月 日

-End-